CLINICAL TRIAL: NCT05468814
Title: Comparison of Two Techniques for the Treatment of Carpal Tunnel Syndrome: A Randomized Clinical Trial
Brief Title: Comparison of Two Techniques for the Treatment of Carpal Tunnel Syndrome
Acronym: STCCOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Irene Calzado Álvarez de Lara, Principal Investigator, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STCOT
Record Dates: First submitted 2022-07-14; First posted 2022-07-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Pillar pain; Grip strength; Pincer strength
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of two treatment groups in a 1:1 ratio, using a computer-generated random assignment list
Who Masked: Participant, Care Provider
Masking Description: This is a double-blind study, in which both the patient and the evaluating staff are unaware of the surgical technique used (both surgeons will perform both techniques). A traumatologist will analyze (before and after surgery) the clinic, strength and satisfaction of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Z-plasty (Experimental): It is a surgical technique in which a Z-shaped section of the transverse carpal ligament is performed, to later join both ends with a resorbable stitch.
  Interventions: Procedure: Z-plasty
- Conventional (Active Comparator): It is a surgical technique in which a complete section of the transverse carpal ligament is performed, without subsequent closure.
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: Z-plasty — It is a surgical technique in which a Z-shaped section of the transverse carpal ligament is performed, to later join both ends with a resorbable stitch.
  Arms: Z-plasty
Procedure: Conventional — It is a surgical technique in which a complete section of the transverse carpal ligament is performed, without subsequent closure.
  Arms: Conventional

SUMMARY:
The main objective of this study is to compare the complete section of the transverse carpal ligament with another median nerve release technique and to determine if the incidence of post-surgical pillar pain is lower for either of the two surgical techniques. As secondary objectives, we also seek to determine if the postsurgical grip and pincer strength and the Boston Carpal Tunnel Questionnaire (BCTQ) score are better for either of the two surgical techniques.

DETAILED DESCRIPTION:
It will be a randomized clinical trial with a sample size of about 80 patients. It will have two study groups: the experimental group (in which 40 patients will be included) where a Z-plasty technique will be applied; and the control group (another 40 patients) who will undergo the conventional technique of complete section of the transverse carpal ligament. The main variable will be the presence or absence of post-surgical pillar pain and, as secondary variables, the recovery of grip and pincer strength and the improvement in the BCTQ score will be studied.

The study population will be patients with carpal tunnel syndrome diagnosed clinically (pain and paresthesias in the first three fingers and radial edge of the fourth finger, nocturnal paresthesias, thenar muscle atrophy, loss of thumb opposition), examination (Durkan's signs , Phalen and Tinnel positive) and with a positive electromyogram test classified as "moderate" or "severe". As inclusion criteria, patients >18 years of age with moderate-severe carpal tunnel syndrome whose symptoms hinder the daily activities of the patient and who have failed conservative treatment will be considered. Those who have already undergone a previous surgical intervention for carpal tunnel syndrome in the same hand, who have traumatic or congenital sequelae in the hand or who do not have the capacity to understand the process or the tests to be performed will be excluded.

The total expected duration of each patient in the study will be 6 months and the following visits and procedures will be carried out: clinical study and quality questionnaires prior to surgery and post-surgical follow-up at 3-4 weeks and at 6 months in consultation, with repetition of clinical examination and quality questionnaires.

The incidence of pillar pain (defined as pain/sensation of allodynia in the area of the thenar and/or hypothenar eminence, hyperalgesia in the scar, pain when supporting the heel of the hand, dysesthesia at rest) will be analyzed applying the principle of intention to treat, using the Mann Whitney test to compare the score in the tests used.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Moderate-severe carpal tunnel syndrome
* Symptoms that hinder the patient's daily activities
* Correct conservative treatment without success

Exclusion Criteria:

* Previous surgical intervention for carpal tunnel syndrome
* Traumatic or congenital sequelae of the hand
* Incompetence to understand the process and the tests to be carried out

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Spain

REFERENCES:
- [Background] Genova A, Dix O, Saefan A, Thakur M, Hassan A. Carpal Tunnel Syndrome: A Review of Literature. Cureus. 2020 Mar 19;12(3):e7333. doi: 10.7759/cureus.7333. PMID 32313774
- [Background] Ludlow KS, Merla JL, Cox JA, Hurst LN. Pillar pain as a postoperative complication of carpal tunnel release: a review of the literature. J Hand Ther. 1997 Oct-Dec;10(4):277-82. doi: 10.1016/s0894-1130(97)80042-7. PMID 9399176
- [Background] Murthy PG, Goljan P, Mendez G, Jacoby SM, Shin EK, Osterman AL. Mini-open versus extended open release for severe carpal tunnel syndrome. Hand (N Y). 2015 Mar;10(1):34-9. doi: 10.1007/s11552-014-9650-x. PMID 25767419
- [Background] Bai J, Kong L, Zhao H, Yu K, Zhang B, Zhang J, Tian D. Carpal tunnel release with a new mini-incision approach versus a conventional approach, a retrospective cohort study. Int J Surg. 2018 Apr;52:105-109. doi: 10.1016/j.ijsu.2018.02.033. Epub 2018 Feb 20. PMID 29471152
- [Background] Khoshnevis J, Layegh H, Yavari N, Eslami G, Afsharfard A, Reza Kalantar-Motamedi SM, Zarrintan S. Comparing open conventional carpal tunnel release with mini-incision technique in the treatment of carpal tunnel syndrome: A non-randomized clinical trial. Ann Med Surg (Lond). 2020 May 16;55:119-123. doi: 10.1016/j.amsu.2020.05.001. eCollection 2020 Jul. PMID 32477509
- [Background] Chen L, Duan X, Huang X, Lv J, Peng K, Xiang Z. Effectiveness and safety of endoscopic versus open carpal tunnel decompression. Arch Orthop Trauma Surg. 2014 Apr;134(4):585-93. doi: 10.1007/s00402-013-1898-z. Epub 2014 Jan 12. PMID 24414237
- [Background] Michelotti BM, Vakharia KT, Romanowsky D, Hauck RM. A Prospective, Randomized Trial Comparing Open and Endoscopic Carpal Tunnel Release Within the Same Patient. Hand (N Y). 2020 May;15(3):322-326. doi: 10.1177/1558944718812129. Epub 2018 Nov 21. PMID 30461319
- [Background] Shin EK. Endoscopic Versus Open Carpal Tunnel Release. Curr Rev Musculoskelet Med. 2019 Dec;12(4):509-514. doi: 10.1007/s12178-019-09584-0. PMID 31773481
- [Background] Kang HJ, Koh IH, Lee TJ, Choi YR. Endoscopic carpal tunnel release is preferred over mini-open despite similar outcome: a randomized trial. Clin Orthop Relat Res. 2013 May;471(5):1548-54. doi: 10.1007/s11999-012-2666-z. Epub 2012 Oct 26. PMID 23100191
- [Background] Hu K, Zhang T, Xu W. Intraindividual comparison between open and endoscopic release in bilateral carpal tunnel syndrome: a meta-analysis of randomized controlled trials. Brain Behav. 2016 Feb 16;6(3):e00439. doi: 10.1002/brb3.439. eCollection 2016 Mar. PMID 27099801
- [Background] Zuo D, Zhou Z, Wang H, Liao Y, Zheng L, Hua Y, Cai Z. Endoscopic versus open carpal tunnel release for idiopathic carpal tunnel syndrome: a meta-analysis of randomized controlled trials. J Orthop Surg Res. 2015 Jan 28;10:12. doi: 10.1186/s13018-014-0148-6. PMID 25627324
- [Background] Orhurhu V, Orman S, Peck J, Urits I, Orhurhu MS, Jones MR, Manchikanti L, Kaye AD, Odonkor C, Hirji S, Cornett EM, Imani F, Varrassi G, Viswanath O. Carpal Tunnel Release Surgery- A Systematic Review of Open and Endoscopic Approaches. Anesth Pain Med. 2020 Dec 26;10(6):e112291. doi: 10.5812/aapm.112291. eCollection 2020 Dec. PMID 34150584
- [Background] Teng X, Xu J, Yuan H, He X, Chen H. Comparison of Wrist Arthroscopy, Small Incision Surgery, and Conventional Surgery for the Treatment of Carpal Tunnel Syndrome: A Retrospective Study at a Single Center. Med Sci Monit. 2019 Jun 3;25:4122-4129. doi: 10.12659/MSM.912912. PMID 31155608
- [Background] Xu L, Huang F, Hou C. Treatment for carpal tunnel syndrome by coronal Z-type lengthening of the transverse carpal ligament. J Pak Med Assoc. 2011 Nov;61(11):1068-71. PMID 22125980
- [Background] Castro-Menendez M, Pagazaurtundua-Gomez S, Pena-Paz S, Huici-Izco R, Rodriguez-Casas N, Montero-Vieites A. Z-Elongation of the transverse carpal ligament vs. complete resection for the treatment of carpal tunnel syndrome. Rev Esp Cir Ortop Traumatol. 2016 Nov-Dec;60(6):355-365. doi: 10.1016/j.recot.2016.06.007. Epub 2016 Aug 25. English, Spanish. PMID 27569033
- [Background] Dias JJ, Bhowal B, Wildin CJ, Thompson JR. Carpal tunnel decompression. Is lengthening of the flexor retinaculum better than simple division? J Hand Surg Br. 2004 Jun;29(3):271-6. doi: 10.1016/j.jhsb.2004.01.011. PMID 15142699
- [Background] Karlsson MK, Lindau T, Hagberg L. Ligament lengthening compared with simple division of the transverse carpal ligament in the open treatment of carpal tunnel syndrome. Scand J Plast Reconstr Surg Hand Surg. 1997 Mar;31(1):65-9. doi: 10.3109/02844319709010507. PMID 9075290
- [Background] Saravi MS, Kariminasab MH, Bari M, Ghaffari S, Razavipour M, Daneshpoor SM, Yazdi MV, Davoudi MM, Azar MS. A Comparison of Hand Pain and Hand Function after Z-plasty Reconstruction of the Transverse Carpal Ligament with Traditional Median Neurolysis in Carpal Tunnel Syndrome. Arch Bone Jt Surg. 2016 Apr;4(2):145-9. PMID 27200393
- [Background] Netscher D, Steadman AK, Thornby J, Cohen V. Temporal changes in grip and pinch strength after open carpal tunnel release and the effect of ligament reconstruction. J Hand Surg Am. 1998 Jan;23(1):48-54. doi: 10.1016/S0363-5023(98)80088-9. PMID 9523954
- [Background] Faour-Martín O, Martín-Ferrero MA, Valverde JA, Zuil-Acosta P, Amigo-Liñares L, Alarcón-García J, De la Red MA. The Simonetta Technique for Carpal Tunnel Syndrome: Immediate Postoperative Evaluation and Long-Term Comparative Study. Int Journal of Orthopaedics. 2014 1(3): 109-115
- [Background] Zhang X, Li Y, Wen S, Zhu H, Shao X, Yu Y. Carpal tunnel release with subneural reconstruction of the transverse carpal ligament compared with isolated open and endoscopic release. Bone Joint J. 2015 Feb;97-B(2):221-8. doi: 10.1302/0301-620X.97B2.34423. PMID 25628286
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not specified. The assignment was randomized
Period: Overall Study
Arm/Group | Z-plasty | Conventional
Started | 60 | 60
Completed | 55 | 54
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Z-plasty | Conventional | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (10.8) | 56.7 (12.7) | 56.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 35 | 80
  Male | 10 | 19 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Laterality [Number; unit: Number of participants right handed] | 29 | 32 | 61
Atrophy [Count of Participants; unit: Participants] | 1 | 2 | 3
Baseline grip strength [Mean (Standard Deviation); unit: kilograms] | 16.3 (8.2) | 19.6 (10.4) | 17.9 (9.5)
Baseline pinch strength [Mean (Standard Deviation); unit: kilograms] | 2.9 (2.2) | 3.9 (2.4) | 3.4 (2.4)
Baseline clinical BCTQ [Mean (Standard Deviation); unit: units on a scale] — Boston Carpal Tunnel Questionnaire. Scale from best to worst (1 - 5)
  units on a scale | 3.5 (0.8) | 3.3 (0.7) | 3.4 (0.8)
Baseline functional BCTQ [Mean (Standard Deviation); unit: units on a scale] — Boston Carpal Tunnel Questionnaire. Scale from best to worst (1 - 5)
  units on a scale | 3.1 (0.9) | 2.8 (0.8) | 3.0 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pillar Pain
Description: Pain/allodynia in the area of the thenar and/or hypothenar eminences, scar hyperalgesia, pain when supporting the heel of the hand, dysesthesia
Time Frame: 3 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
Participants | 14 | 24

2. Primary Outcome: Incidence of Pillar Pain
Description: as for outcome 1
Time Frame: 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
Participants | 5 | 9

3. Secondary Outcome: Grip Strength
Description: Grip strength measured with a dynamometer
Time Frame: 3 weeks after surgery
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
kilograms | 13.8 (7.0) | 15.6 (9.5)

4. Secondary Outcome: Grip Strength
Description: Grip strength measured with a dynamometer
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
kilograms | 18.6 (8.9) | 19.1 (9.0)

5. Secondary Outcome: Pinch Strength
Description: Pinch strength measured with a dynamometer
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
kilograms | 3.8 (2.8) | 3.5 (2.5)

6. Secondary Outcome: Pinch Strength
Description: Pinch strength measured with a dynamometer
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
kilograms | 5.4 (3.0) | 5.1 (2.4)

7. Secondary Outcome: Clinical BCTQ
Description: Boston Carpal Tunnel Syndrome Questionnaire used to evaluate the clinic of carpal tunnel syndrome.
  Minimum: 1 (better). Maximum: 5 (worse)
Time Frame: 3 weeks after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
units on a scale | 1.9 (0.8) | 1.8 (0.7)

8. Secondary Outcome: Functional BCTQ
Description: as for outcome 7
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
units on a scale | 1.7 (0.8) | 1.6 (0.7)

9. Secondary Outcome: Clinical BCTQ
Description: Boston Carpal Tunnel Syndrome Questionnaire used to evaluate the clinic (symptoms) of carpal tunnel syndrome.
  Minimum: 1 (better). Maximum: 5 (worse)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
units on a scale | 1.5 (0.8) | 1.5 (0.7)

10. Secondary Outcome: Functional BCTQ
Description: Boston Carpal Tunnel Syndrome Questionnaire used to evaluate the clinic (functionality; daily activities) of carpal tunnel syndrome.
  Minimum: 1 (better). Maximum: 5 (worse)
Time Frame: 3 weeks after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Z-plasty | Conventional
Number analyzed (Participants) | 55 | 54
units on a scale | 2.2 (0.9) | 2.1 (0.8)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Major surgical complications: infection, wound dehiscence, amputation...
Arm/Group | Z-plasty | Conventional
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT05468814/Prot_SAP_000.pdf